CLINICAL TRIAL: NCT06535633
Title: Community-based Exercise for Older Adults With Chronic Musculoskeletal Pain: a Randomised Controlled Feasibility Trial
Brief Title: Community-based Exercise for Older Adults With Chronic Musculoskeletal Pain
Acronym: ComEx Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024_02_23_EHS; DIFA-2-23-024, 7272 (Other: Health Research Board)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: chronic musculoskeletal pain,; exercise; feasibility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm: Exercise classes (Experimental): The investigators have trained exercise trainers in Pain neuroscience and they will lead a set of classes, adapted to the needs of people with chronic pain. Focus groups with people with chronic pain detailed the important factors to consider in planning an exercise intervention, these being that the activity should be enjoyable, non-competitive and accessible to all levels of physical activity, and the venues should offer easy access with public transport. The investigators have identified three exercise types from the current LSP offerings that could meet the needs of people with chronic MSK pain, namely Tai Chi, Activator Pole walking and Aquarobics, which will run once a week for 8 weeks. The intervention group will also receive a paper-based education manual about physical activity and pain management education designed for people with chronic pain.
  Interventions: Other: Intervention arm: Exercise class
- Control (No Intervention): The control group comprises the same paper-based education manual about physical activity and pain management education designed for people with chronic pain and based on the "Explain Pain" principles. These participants will continue with usual care for their chronic pain. Based on PPI feedback suggesting the importance of equity for all who volunteer to take part, those in the control group will be offered the opportunity to participate in the intervention (group exercise classes) after they have completed their final follow up assessments.

INTERVENTIONS:
Other: Intervention arm: Exercise class — The exercise trainers, who are educated in chronic pain, will lead a set of classes, adapted to the needs of people with chronic pain. The investigators have conducted PPI activities with the members of Chronic Pain Ireland, to understand the barriers and facilitators for community-based exercise and their needs in relation to same. A forthcoming publication reports the results of a survey of a survey of (n=130) members of CPI highlightinged that key barriers to community-based exercise included fear of pain exacerbation, and not having skilled exercise instruction. The exercise modalities of choice have been informed by the survey results as well as alignment with the LSP class offerings and trainer competency. Classes on offer are focused on aquatic exercise, Activator pole walking, yoga or Pilates, and circuit-style fitness, for participants to choose their own preferred option. Classes will run weekly for 8 weeks, duration 1 hour.
  Arms: Intervention arm: Exercise classes

SUMMARY:
Chronic pain management services in Ireland are severely under-resourced. There is a key opportunity for community-based exercise to address some of the needs of people early in their chronic pain journey and potentially prevent or reduce their needs for secondary healthcare support, reducing the burden on healthcare waiting lists.

Musculoskeletal pain is a significant barrier to participation in physical activity for these older adults, and at present, community-based exercise trainers do not have any education or resources to help support people with chronic pain to sustain their participation in physical activity programmes. Healthcare professionals who hold negative beliefs in relation to the role of physical activity for chronic pain are more likely to provide advice that reinforces unhelpful behaviours and increases disability. Pain education has been shown to positively change beliefs and shift views towards more evidence-based physical activity recommendations in a range of professionals including physiotherapists, nurses and sports therapists. In addition, specific psychological and behavioural approaches to support self-efficacy, develop pacing skills, and manage pain flareups are required to help people with chronic pain sustain their engagement in exercise. Appropriate education is required to equip those working with people in chronic pain to facilitate these skills. While exercise is a safe intervention, there are key differences in how people with chronic pain may respond to or recover from exercise that need to be planned for in exercise programmes. People with chronic pain vary greatly in their abilities and functional limitations, goals, and lifestyle, in comparison to those without troublesome pain. A review of qualitative data from people with fibromyalgia showed that they report self-selecting an exercise intensity lower than the guideline recommended level to avoid adverse effects and build pain management skills. Patient-public involvement (PPI) focus groups and a survey conducted in the development of this protocol showed that people with chronic pain were very reluctant to enrol in current community-based physical activity opportunities due to anxiety that the exercise leader would not understand or be able to meet their specific needs, and the consequent fear of symptom exacerbation. The most important priority identified for their participation was having an exercise leader who was trained in supporting people with pain. Exercise that is tailored to the specific needs of people with pain is likely to offer a more supportive, safe, and effective approach. There is a clear need for a project developing and delivering an educational intervention for exercise trainers, to support people with pain to exercise in their community.

DETAILED DESCRIPTION:
The investigators have trained exercise trainers in Pain neuroscience and they will lead a set of classes, adapted to the needs of people with chronic pain. In addition, the investigators have conducted PPI activities with the members of Chronic Pain Ireland, to understand the barriers and facilitators for community-based exercise and their needs in relation to same. A survey of (n=130) members of CPI highlighted key barriers to community-based exercise included fear of pain exacerbation, and not having a skilled exercise leader. Access to an exercise trainer trained in supporting people with chronic pain was the top facilitator of engagement with exercise chosen by respondents. Focus groups with people with chronic pain detailed the important factors to consider in planning an exercise intervention, these being that the activity should be enjoyable, non-competitive and accessible to all levels of physical activity, and the venues should offer easy access with public transport. Based on this data and framed within the biopsychosocial model of chronic pain (Figure 1), a number of exercise types from the current LSP offerings that could meet the needs of people with chronic MSK pain, namely Tai Chi, Activator Pole walking and Aquarobics were identified. These classes run once a week for 8 weeks. The intervention group will also receive a paper-based education manual about physical activity and pain management education designed for people with chronic pain and based on the "Explain Pain" principles.

The control group comprises the same paper-based education manual about physical activity and pain management education designed for people with chronic pain and based on the "Explain Pain" principles. These participants will continue with usual care for their chronic pain. Based on PPI feedback suggesting the importance of equity for all who volunteer to take part, those in the control group will be offered the opportunity to participate in the intervention (group exercise classes) after they have completed their final follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be aged 50 or older,
* report chronic MSK pain of ≥3 months duration,
* not currently meeting the exercise guidelines of 150 minutes of moderate physical activity per week (determined using the International Physical Activity Questionnaire (IPAQ)

Exclusion Criteria:

* Participants will be excluded if they have health conditions which could be worsened by exercise (e.g. neurological, or cardiovascular conditions, post-exertional malaise (screened using the DePaul Post-Exertional Malaise Questionnaire have recently undergone trauma or surgery, or have significant mobility issues which would limit exercise participation.
* Participants who are unable to communicate in English sufficiently to complete consent or baseline assessment will be excluded

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 2 month periods
  Overall numbers recruited per month during the recruitment phases
Retention rate | End of intervention 8 weeks post baseline assessment
  Retention will be defined as the proportion of participants who complete baseline and post intervention measures.
Refusal rate | 2 month periods of recruitment
  • Refusal rate will be recorded as the number of eligible individuals who are invited to partake in the study but refuse to do so, with reasons recorded
Attendance rates at classes | each class for eight weeks
  • Attendance rates at classes will be reported as mean % attendance rates at classes, as well as the proportion of participants attending a minimum of 60% of classes (via attendance log taken at exercise classes) as the minimum acceptable attendance level.

SECONDARY OUTCOMES:
Pain Numerical Rating Scale for average pain intensity | Baseline
  Pain intensity will be measured as average pain for the previous week, using a 0-10 Numerical Rating Scale (NRS). The NRS has been shown to have acceptable reliability and validity in a range of chronic pain population
Pain Numerical Rating Scale for average pain intensity | End of intervention and corresponding control period: 8 weeks
  Pain intensity will be measured as average pain for the previous week, using a 0-10 Numerical Rating Scale (NRS). The NRS has been shown to have acceptable reliability and validity in a range of chronic pain population
Function via The Pain Disability Index (PDI) | Baseline
  The Pain Disability Index (PDI) is a 7-item questionnaire to investigate the magnitude of self-reported pain-related disability, independent from region of pain or pain-related diagnosis. The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability. The sum of the seven items equals the total score of the PDI, which ranges from 0 to 70, with higher scores reflecting higher interference of pain with daily activities. It has been widely validated in populations with chronic musculoskeletal pain
Function via The Pain Disability Index (PDI) | End of intervention and corresponding control period: 8 weeks
  The Pain Disability Index (PDI) is a 7-item questionnaire to investigate the magnitude of self-reported pain-related disability, independent from region of pain or pain-related diagnosis. The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability. The sum of the seven items equals the total score of the PDI, which ranges from 0 to 70, with higher scores reflecting higher interference of pain with daily activities. It has been widely validated in populations with chronic musculoskeletal pain
Emotional function: Hospital Anxiety and Depression Scale (HADS) | Baseline
  Emotional function: Hospital Anxiety and Depression Scale The HADS was originally a 14-item questionnaire to assess levels of depression and anxiety in hospital patients. It has been widely used in chronic pain research, but a recent factor analysis involving over 2500 people with chronic MSK pain showed that an 11-item version was a more valid and reliable measure of emotional distress related to pain than the full instrument, therefore the 11-item version will be used in the feasibility study. The results suggested that an 11-item refined version of the HADS could be considered as a unidimensional scale and, if implemented, could be suitable for the measurement of emotional distress in this population.
  Minimum value: 0, maximum value: 11. Higher value indicates greater emotional distress
Emotional function: Hospital Anxiety and Depression Scale (HADS) | End of intervention and corresponding control period: 8 weeks
  The HADS was originally a 14-item questionnaire to assess levels of depression and anxiety in hospital patients. It has been widely used in chronic pain research, but a recent factor analysis involving over 2500 people with chronic MSK pain showed that an 11-item version was a more valid and reliable measure of emotional distress related to pain than the full instrument, therefore the 11-item version will be used in the feasibility study.
  Minimum value: 0, maximum value: 11. Higher value indicates greater emotional distress
Rating of satisfaction/improvement | Baseline
  Rating overall improvement has been recommended as a core outcome in chronic pain, therefore a Global Rating of Change score is included, designed to quantify a participant's improvement or deterioration over time (Bobos et al. 2020). This is a 7 numbered scale balanced in the centre with "unchanged", and anchored with "very much worse" on the left, and "completely recovered" on the right" and the following prompt: With respect to your pain problem, how would you describe yourself now compared to when you began the study?.
  The patient responds to the question by marking a scale that measures the degree of improvement or deterioration. The midpoint is important so that the patient is not forced to rate himself or herself as better or worse in the event that the condition has remained the same.
  Minimum value: 1, maximum value:7, greater scores indicate a positive satisfaction response
Rating of satisfaction/improvement | End of intervention and corresponding control period: 8 weeks
  Rating overall improvement has been recommended as a core outcome in chronic pain, therefore a Global Rating of Change score, designed to quantify a participant's improvement or deterioration over time, will be used. This is a 7 numbered scale balanced in the centre with "unchanged", and anchored with "very much worse" on the left, and "completely recovered" on the right" and the following prompt: With respect to your pain problem, how would you describe yourself now compared to when you began the study? The patient responds to the question by marking a scale that measures the degree of improvement or deterioration. The midpoint is important so that the patient is not forced to rate himself or herself as better or worse in the event that the condition has remained the same.
  Minimum value: 1, maximum value:7, greater scores indicate a positive satisfaction response
Physical activity objective via accelerometry | 7 days at baseline
  ActivPAL : Time spent in sedentary and non sedentary activity will be measured using the ActivPAL™ (PAL Technologies Ltd, Glasgow, UK). The ActivPAL™ is a small, lightweight activity monitor that classifies an individual's free-living activity into time periods spent in sedentary, standing and walking positions using proprietary algorithms.
  The ActivPAL™ is a uni-axial accelerometer which produces a signal related to thigh inclination. The ActivPAL™ also records step count, i.e. number of steps taken, and transition count, i.e. number of movements from lying/sitting positions to standing and vice versa. The ActivPAL™ will be worn for 7 days at baseline and 7 days after the completion of the exercise intervention.
Physical activity objective | 7 days after completion of the exercise intervention
  ActivPAL ActivPAL : Time spent in sedentary and non sedentary activity will be measured using the ActivPAL™ (PAL Technologies Ltd, Glasgow, UK). The ActivPAL™ is a small, lightweight activity monitor that classifies an individual's free-living activity into time periods spent in sedentary, standing and walking positions using proprietary algorithms.
  The ActivPAL™ is a uni-axial accelerometer which produces a signal related to thigh inclination. The ActivPAL™ also records step count, i.e. number of steps taken, and transition count, i.e. number of movements from lying/sitting positions to standing and vice versa. The ActivPAL™ will be worn for 7 days at baseline and 7 days after the completion of the exercise intervention.
Physical activity subjective via International Physical Activity Questionnaire | Baseline
  International Physical Activity Questionnaire (IPAQ) which measures duration and frequency of physical activity over the preceding 7 days across a range of domains including leisure time, domestic and gardening activities, work-related and transport-related activity, and has been shown to be reliable in populations with chronic MSK conditions.
  Scoring categories:
  Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
  Scoring a MODERATE level of physical activity on the IPAQ means you are doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.
Physical activity subjective via International Physical Activity Questionnaire | End of intervention and corresponding control period: 8 weeks
  International Physical Activity Questionnaire (IPAQ) which measures duration and frequency of physical activity over the preceding 7 days across a range of domains including leisure time, domestic and gardening activities, work-related and transport-related activity, and has been shown to be reliable in populations with chronic MSK conditions.
  Scoring categories:
  Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level.
  Scoring a MODERATE level of physical activity on the IPAQ means you are doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days.
  Scoring a LOW level of physical activity on the IPAQ means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.
Health-related quality of life via EQ-5d-5l,( EuroQol) | Baseline
  The EQ-5d-5l, a valid and response measure of health-related quality of life, covering five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension in the descriptive system has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Health-related quality of life | End of intervention and corresponding control period: 8 weeks
  The EQ-5d-5l, a valid and response measure of health-related quality of life, covering five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension in the descriptive system has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Karen McCreesh, PhD, Principal Investigator — UL
Locations (1):
- University of Limerick, Ireland, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analysed during the current study and will be available upon request from Dr Mairéad Conneely, mairead.c.conneely@ul.ie
Supporting Information: Study Protocol, SAP
Time Frame: Once the protocol is published, it will be shared and available on the published platform.
Access Criteria: Open access